CLINICAL TRIAL: NCT03336333
Title: An International, Phase 3, Open-Label, Randomized Study of BGB-3111 Compared With Bendamustine Plus Rituximab in Patients With Previously Untreated Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma (CLL/SLL)
Brief Title: A Study Comparing Zanubrutinib With Bendamustine Plus Rituximab in Participants With Previously Untreated CLL or SLL
Acronym: SEQUOIA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-304; 2017-001551-31 (EudraCT Number); CTR20190416 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2017-11-01; First posted 2017-11-08 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: zanubrutinib; BTK inhibitor; bendamustine; rituximab; venetoclax; BGB-3111; Phase 3
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib; Bendamustine Hydrochloride; Rituximab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: Bendamustine + Rituximab (Experimental): Participants will receive bendamustine plus rituximab for up to six 28-day cycles (Arm B)
  Interventions: Drug: Bendamustine; Drug: Rituximab
- Cohort 1: Zanubrutinib (Experimental): Participants will receive zanubrutinib until unacceptable toxicity or disease progression (Arm A)
  Interventions: Drug: Zanubrutinib
- Cohort 1a (China only): Bendamustine + Rituximab (Experimental): Participants will receive bendamustine plus rituximab for up to six 28-day cycles (Arm B, China only)
  Interventions: Drug: Bendamustine; Drug: Rituximab
- Cohort 1a (China only): Zanubrutinib (Experimental): Participants will receive zanubrutinib until unacceptable toxicity or disease progression (Arm A, China only)
  Interventions: Drug: Zanubrutinib
- Cohort 2: Zanubrutinib (Experimental): Participants will receive zanubrutinib until unacceptable toxicity or disease progression (Arm C)
  Interventions: Drug: Zanubrutinib
- Cohort 3: Venetoclax + Zanubrutinib (Experimental): Approximately 110 participants, 50 without del17p and 60 with del[17p] or TP53 mutation will receive zanubrutinib plus venetoclax; Participants will also receive zanubrutinib starting on Cycle 1 Day 1 then daily for a minimum of 27 cycles, or until unacceptable toxicity or disease progression, whichever occurs first. Participants will receive venetoclax starting Cycle 4 Day 1 according to a 5-week dose-up schedule then daily until unacceptable toxicity, disease progression, or for a maximum of 24 cycles. Each cycle is 28 days. (Arm D)
  Interventions: Drug: Zanubrutinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Zanubrutinib — Administered as two 80-milligram (mg) capsules by mouth twice a day (160 mg twice a day)
  Other Names: BGB-3111; BRUKINSA
  Arms: Cohort 1: Zanubrutinib; Cohort 1a (China only): Zanubrutinib; Cohort 2: Zanubrutinib; Cohort 3: Venetoclax + Zanubrutinib
Drug: Bendamustine — Administered intravenously (IV) at a dose of 90 mg/m^2/day on the first 2 days of each cycle for 6 cycles.
  Other Names: Treanda, Ribomustin, and Levact
  Arms: Cohort 1: Bendamustine + Rituximab; Cohort 1a (China only): Bendamustine + Rituximab
Drug: Rituximab — Administered intravenously (IV) at a dose of 375 mg/m^2 on day 0 of cycle 1, and at a dose of 500 mg/m^2 on day 1 of cycles 2 to 6
  Other Names: Rituxan, MabThera
  Arms: Cohort 1: Bendamustine + Rituximab; Cohort 1a (China only): Bendamustine + Rituximab
Drug: Venetoclax — 400 mg tablets administered orally once daily.
  Other Names: Venclexta, Venclyxto
  Arms: Cohort 3: Venetoclax + Zanubrutinib

SUMMARY:
To compare efficacy between zanubrutinib versus bendamustine and rituximab in patients with previously untreated CLL/SLL, as measured by progression free survival assess by Independent Central Review.

DETAILED DESCRIPTION:
This is a global phase 3, open label, randomized study of zanubrutinib versus bendamustine plus rituximab (B+R) in participants with previously untreated chronic lymphocytic leukemia or small lymphocytic lymphoma (CLL/SLL), including participants without del(17p) [Cohort 1] and participants with del(17p) [Cohort 2 and Cohort 3]. Participants in Cohort 1 are randomized 1:1 to zanubrutinib (Arm A) or bendamustine plus rituximab (Arm B). Randomization will be stratified by age, Binet stage, immunoglobulin variable region heavy chain (IGHV) mutational status, and geographic region. Participants in Cohort 2 will receive treatment with zanubrutinib. Participants in Cohort 3 will receive treatment with zanubrutinib and venetoclax.

ELIGIBILITY:
Key Inclusion Criteria:

* Unsuitable for chemoimmunotherapy with fludarabine, cyclophosphamide, and rituximab (FCR)
* Confirmed diagnosis of CD20-positive CLL or SLL, requiring treatment
* Measurable disease by imaging
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Life expectancy ≥ 6 months
* Adequate bone marrow function
* Adequate renal and hepatic function

Key Exclusion Criteria:

* Previous systemic treatment for CLL/SLL
* Requires ongoing need for corticosteroid treatment
* Known prolymphocytic leukemia or history of or suspected Richter's transformation.
* Clinically significant cardiovascular disease
* Prior malignancy within the past 3 years, except for curatively treated basal or squamous cell skin cancer, non-muscle-invasive bladder cancer, carcinoma in situ of the cervix of breast, or localized Gleason score 6 prostate cancer
* History of severe bleeding disorder
* History of stroke or intracranial hemorrhage within 6 months before the first dose of study drug
* Severe or debilitating pulmonary disease
* Inability to swallow capsules or disease affecting gastrointestinal function
* Active infection requiring systemic treatment
* Known central nervous system involvement by leukemia or lymphoma
* Underlying medical condition that will render the administration of study drug hazardous or obscure interpretation of toxicity or AEs
* Known infection with human immunodeficiency virus (HIV) or active hepatitis B or C infection
* Major surgery ≤ 4 weeks prior to start of study treatment
* Pregnant or nursing females
* Vaccination with live vaccine within 35 days prior to the first dose of study drug.
* Ongoing alcohol or drug addiction
* Known hypersensitivity to zanubrutinib, bendamustine, rituximab, or venetoclax (as applicable) or any other ingredients of the study drugs
* Requires ongoing treatment with strong cytochrome P450 (CYP3A) inhibitor or inducer
* Concurrent participation in another therapeutic clinical study

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2026-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (158):
- United States (18):
  - Augusta University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Research Medical Center, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Summit Medical Group, Florham Park, New Jersey
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Prairie Lakes Healthcare System, Watertown, South Dakota
  - Tennessee Oncology, Pllc Nashville, Nashville, Tennessee
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - University of Virginia, Charlottesville, Virginia
  - Va Puget Sound Health Care System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (16):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - The Tweed Valley Hospital, Cudgen, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Centre Wesley, Auchenflower, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Peninsula Private Hospital, Frankston, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (5):
  - Medizinische Universitatsklinik Innsbruck, Innsbruck
  - Krankenhaus Der Barmherzigen Schwestern Linz, Linz
  - Allgemeines Krankenhaus Der Stadt Linz, Linz
  - Universitatsklinik Fur Innere Medizin Iii Universitatsklinikum Der Pmu Landeskrankenhaus Salzburg, Salzburg
  - Klinikum Wels Grieskirchen, Wels
- Belgium (5):
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Universitaire (Chu) de Liege Site Du Sart Tilman, Liège
  - Clinique Saint Pierre, Ottignies
  - Centre Hospitalier Universitaire Universite Catholique de Louvain Site Godinne, Yvoir
- China (19):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Second Affiliated Hospital of Army Medical University (Xinqiao Hospital), Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Quanzhou First Affliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University Branch Shizi, Suzhou, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Czechia (4):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Olomouc, Olomouc
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- France (17):
  - Centre Hospitalier Victor Dupouy Dargenteuil, Argenteuil
  - Centre de Lutte Contre Le Cancer Institut Bergonie, Bordeaux
  - Chu Caen Normandie, Caen
  - Centre Hospitalier Departemental de Vendee, La Roche-sur-Yon
  - Centre Hospitalier Le Mans, Le Mans
  - Centre Hospitalier Universitaire Limoges Chu de Limoges, Limoges
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier Universitaire Nantes Hotel Dieu, Nantes
  - Hopital de La Pitie Salpetriere, Paris
  - Groupe Hospitalier Du Haut Leveque, Pessac
  - Chu Hopital Lyon Sud, PierreBenite
  - Centre Hospitalier Universitaire de Poitier Hopital de La Miletrie Hopital Jean Bernard, Poitiers
  - Hopital Robert Debre, Reims
  - Hopital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Chu Tours Hopital Bretonneau Service Pneumologie, Tours
  - Chu Nancy Hopital Brabois, VandoeuvrelesNancy
- Italy (11):
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori Irst, Meldola
  - Fondazione Irccs Ca Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Universita Degli Studi Di Modena Azienda Ospedaliere Policlinco, Modena
  - Azienda Unita Sanitaria Locale Di Ravenna, Ravenna
  - Universita Degli Studi La Sapienza, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera S Maria Di Terni, Terni
  - Ao Citta Della Salute E Della Scienza Di Torino Presidio O, Torino
- New Zealand (5):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Palmerston North Hospital, Palmerston North
  - North Shore Hospital, Takapuna
  - Tauranga Hospital, Tauranga
- Poland (9):
  - Szpital Specjalist W Brzozowie,Podkarpacki Osrodek Onkologiczny, Brzozów
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Chorzów
  - Copernicus Podmiot Leczniczy Sp Z Oo Wojewodzkie Centrum Onkologii, Gdansk
  - Szpitale Pomorskie Spolka Z Ograniczona Odpowiedzialnoscia, Gdynia
  - Centrum Onkologii Instytut Im Marii Sklodowskiej Curie, Oddzial W Gliwicach, Gliwice
  - Malopolskie Centrum Medyczne Sc, Krakow
  - Wojewodzki Szpital Specjalistyczny W Legnicy, Legnica
  - Wielospecjalistyczne Centrum Onkologii I Traumatologii Im M Kopernika W Lodzi, Lodz
  - Centrum Onkologii Ziemi Lubelskiej, Lublin
- Russia (15):
  - Kaluga Regional Hospital, Kaluga, Kaluga Oblast
  - State Healthcare Institution Oncologic Dispensary No Health Department of Krasnodar Region, Sochi, Krasnodarskiy Kray
  - N N Blokhin Russian Cancer Research Center Konstantin Laktionov, Moscow, Moscow
  - Russian Academy of Advanced Medical Studies, City Clinical Hospital, Moscow, Moscow
  - Nizhniy Novgorod Regional Clinical Hospital Nasemashko, Nizhny Novgorod, Nizhny Novgorod Oblast
  - State Budgetary Healthcare Institution Regional Clinical Dispensary, Penza, Penza Oblast
  - State Budgetary Healthcare Institution of Perm Krai Clinical Medical Sanitary Establishment, Perm, Permskiy Kray
  - Kemerovo Regional Clinical Hospital Na Sv Belyaev, Kemerovo, Pskov Oblast
  - Ryazan Regional Clinical Hospital, Ryazan, Ryazan Oblast
  - Fgu Russian Scientific Research Institute of Hematology and Transfusiology, Saint Petersburg, Sankt-Peterburg
  - Sverdlovsk Regional Clinical Hospital, Yekaterinburg, Sverdlovsk Oblast
  - Central City Hospital, Yekaterinburg, Sverdlovsk Oblast
  - Clinical Oncology Dispensary, Kazan, Tambov Oblast
  - Tula Area Clinical Hospital, Tula, Tula Oblast
  - State Budgetary Healthcare Institution Volgograd Regional Clinical Oncology Dispensary, Volgograd, Volgograd Oblast
- Spain (9):
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital Del Mar, Barcelona
  - Institut Catala Doncologia, Barcelona
  - Hospital de La Princesa, Madrid
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Clinica Universidad de Navarra Pamplona, Pamplona
  - Hospital Universitari I Politecnic La Fe, Valencia
  - Hospital de Dia Quironsalud Zaragoza, Zaragoza
- Sweden (6):
  - Medicinkliniken, Borås
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skanes Universitetssjukhus I Lund, Lund
  - Universitetssjukhuset Orebro, Örebro
  - Karolinska Universitetssjukhuset Solna, Stockholm
  - Uppsala Akademiska Sjukhus, Uppsala
- Taiwan (3):
  - Hualien Tzu Chi Hospital, Hualien City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - National Taiwan University Hospital East Campus, Taipei
- United Kingdom (16):
  - Birmingham Heartlands Hospital, Birmingham
  - The Royal Bournemouth and Christchurch Hospitals Nhs Foundation, Bournemouth
  - Cambridge University Hospitals Nhs Foundation Trust, Cambridge
  - Kent and Canterbury Hospital, Canterbury
  - The Christie Hospital, Greater Manchester
  - The Leeds Teaching Hospitals Nhs Trust, Leeds
  - Barts and the London Nhs Trust, London
  - Royal Marsden Hospital, London
  - Sarah Cannon Research Institute Uk, London
  - Maidstone and Tunbridge Wells Nhs Trust, Kent Oncology Centre, Maidstone Hospital, Maidstone
  - Norfolk and Norwich University Hospitals Nhs Foundation Trust, Norwich
  - Nottingham University Hospitals Nhs Trust, Nottingham
  - Derriford Hospital, Plymouth
  - Southampton General Hospital, Southampton
  - Sunderland Royal Hospital, Sunderland
  - The Royal Wolverhampton Nhs Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

REFERENCES:
- [Result] Mu S, Tang Z, Novotny W, Tawashi M, Li TK, Ou Y, Sahasranaman S. Effect of rifampin and itraconazole on the pharmacokinetics of zanubrutinib (a Bruton's tyrosine kinase inhibitor) in Asian and non-Asian healthy subjects. Cancer Chemother Pharmacol. 2020 Feb;85(2):391-399. doi: 10.1007/s00280-019-04015-w. Epub 2019 Dec 26. PMID 31875923
- [Result] Tam CS, Robak T, Ghia P, Kahl BS, Walker P, Janowski W, Simpson D, Shadman M, Ganly PS, Laurenti L, Opat S, Tani M, Ciepluch H, Verner E, Simkovic M, Osterborg A, Trneny M, Tedeschi A, Paik JC, Kuwahara SB, Feng S, Ramakrishnan V, Cohen A, Huang J, Hillmen P, Brown JR. Zanubrutinib monotherapy for patients with treatment naive chronic lymphocytic leukemia and 17p deletion. Haematologica. 2021 Sep 1;106(9):2354-2363. doi: 10.3324/haematol.2020.259432. PMID 33054121
- [Derived] Munir T, Martinez-Calle N, Xu S, Yang K, Ge X, Ali AK, Mohseninejad L, Dobi B, Rakonczai P, Ma H, Williams R, Aldairy W, Lamanna N. Indirect Comparisons of the Efficacy and Safety of Zanubrutinib versus Venetoclax plus Obinutuzumab in Treatment-Naive Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma. Oncol Ther. 2025 Dec;13(4):1055-1070. doi: 10.1007/s40487-025-00380-0. Epub 2025 Sep 13. PMID 40944848
- [Derived] Shadman M, Munir T, Ma S, Lasica M, Tani M, Robak T, Flinn IW, Brown JR, Ghia P, Ferrant E, Tam CS, Janowski W, Jurczak W, Xu L, Tian T, Lefebure M, Agresti S, Hirata J, Tedeschi A. Zanubrutinib and Venetoclax for Patients With Treatment-Naive Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma With and Without Del(17p)/TP53 Mutation: SEQUOIA Arm D Results. J Clin Oncol. 2025 Jul 20;43(21):2409-2417. doi: 10.1200/JCO-25-00758. Epub 2025 May 31. PMID 40448577
- [Derived] Shadman M, Munir T, Robak T, Brown JR, Kahl BS, Ghia P, Giannopoulos K, Simkovic M, Osterborg A, Laurenti L, Walker PA, Opat SS, Ciepluch H, Greil R, Hanna M, Tani M, Trneny M, Brander D, Flinn IW, Grosicki S, Verner E, Tedeschi A, de Guibert S, Tumyan G, Laribi K, Garcia-Marco JA, Li JY, Tian T, Liu Y, Korolkiewicz R, Szeto A, Tam CS, Jurczak W. Zanubrutinib Versus Bendamustine and Rituximab in Patients With Treatment-Naive Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma: Median 5-Year Follow-Up of SEQUOIA. J Clin Oncol. 2025 Mar;43(7):780-787. doi: 10.1200/JCO-24-02265. Epub 2024 Dec 8. PMID 39647999
- [Derived] Kittai AS, Allan JN, James D, Bridge H, Miranda M, Yong ASM, Fam F, Roos J, Shetty V, Skarbnik A, Davids MS. An indirect comparison of acalabrutinib with and without obinutuzumab vs zanubrutinib in treatment-naive CLL. Blood Adv. 2024 Jun 11;8(11):2861-2869. doi: 10.1182/bloodadvances.2023012142. PMID 38598745
- [Derived] Moslehi JJ, Furman RR, Tam CS, Salem JE, Flowers CR, Cohen A, Zhang M, Zhang J, Chen L, Ma H, Brown JR. Cardiovascular events reported in patients with B-cell malignancies treated with zanubrutinib. Blood Adv. 2024 May 28;8(10):2478-2490. doi: 10.1182/bloodadvances.2023011641. PMID 38502198
- [Derived] Ghia P, Barnes G, Yang K, Tam CS, Robak T, Brown JR, Kahl BS, Tian T, Szeto A, Paik JC, Shadman M. Health-related quality-of-life in treatment-naive CLL/SLL patients treated with zanubrutinib versus bendamustine plus rituximab. Curr Med Res Opin. 2023 Nov;39(11):1505-1511. doi: 10.1080/03007995.2023.2262381. Epub 2023 Oct 12. PMID 37752878
- [Derived] Tam CS, Brown JR, Kahl BS, Ghia P, Giannopoulos K, Jurczak W, Simkovic M, Shadman M, Osterborg A, Laurenti L, Walker P, Opat S, Chan H, Ciepluch H, Greil R, Tani M, Trneny M, Brander DM, Flinn IW, Grosicki S, Verner E, Tedeschi A, Li J, Tian T, Zhou L, Marimpietri C, Paik JC, Cohen A, Huang J, Robak T, Hillmen P. Zanubrutinib versus bendamustine and rituximab in untreated chronic lymphocytic leukaemia and small lymphocytic lymphoma (SEQUOIA): a randomised, controlled, phase 3 trial. Lancet Oncol. 2022 Aug;23(8):1031-1043. doi: 10.1016/S1470-2045(22)00293-5. Epub 2022 Jul 7. PMID 35810754

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Available data are presented as of the primary analysis data cut-off date of 07MAY2021; as of the data cut-off date, all cohorts were ongoing.
Groups:
- Cohort 1: Bendamustine + Rituximab Without Del(17p): Bendamustine + rituximab in participants with chronic lymphocytic leukemia (CLL) without deletion 17p [del(17p)]; bendamustine 90 milligrams (mg)/m^2/day administered intravenously (IV) on the first 2 days of each cycle for 6 cycles; rituximab 375 mg/m^2 for Cycle 1 and 500 mg/m^2 for Cycles 2 to 6 (each cycle is 28 days)
- Cohort 1: Zanubrutinib Without Del(17p): Zanubrutinib in participants with CLL without del(17p); 160 mg administered twice a day orally until unacceptable toxicity or disease progression
- Cohort 2: Zanubrutinib With Del(17p): Zanubrutinib in participants with CLL with del(17p); 160 mg administered twice a day orally until unacceptable toxicity or disease progression
Period: Overall Study
Arm/Group | Cohort 1: Bendamustine + Rituximab Without Del(17p) | Cohort 1: Zanubrutinib Without Del(17p) | Cohort 2: Zanubrutinib With Del(17p)
Started | 238 | 241 | 111
Treated | 227 | 240 | 111
Completed | 0 | 0 | 0
Not Completed | 238 | 241 | 111
Not completed — Remained on study at time of data cut-off | 202 | 219 | 102
Not completed — Death | 14 | 16 | 8
Not completed — Withdrawal by Subject | 16 | 5 | 1
Not completed — Physician Decision | 5 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat analysis set included all enrolled participants who were assigned to a treatment group (as of cut-off date of 07MAY2021)
Groups:
- Cohort 1: Bendamustine + Rituximab Without Del(17p): Bendamustine + Rituximab in participants with CLL without del(17p); bendamustine 90 milligrams (mg)/m^2/day administered intravenously (IV) on the first 2 days of each cycle for 6 cycles; rituximab 375 mg/m^2 for Cycle 1 and 500 mg/m^2 for Cycles 2 to 6 (each cycle is 28 days)
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Bendamustine + Rituximab Without Del(17p) | Cohort 1: Zanubrutinib Without Del(17p) | Cohort 2: Zanubrutinib With Del(17p) | Total
Number analyzed (Participants) | 238 | 241 | 111 | 590
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 46 | 45 | 16 | 107
  >=65 years | 192 | 196 | 95 | 483
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 87 | 32 | 213
  Male | 144 | 154 | 79 | 377
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 1 | 10
  Not Hispanic or Latino | 211 | 218 | 99 | 528
  Unknown or Not Reported | 23 | 18 | 11 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 9 | 4 | 1 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 1 | 4 | 0 | 5
  White | 206 | 221 | 105 | 532
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 22 | 11 | 5 | 38

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Progression-free Survival (PFS) as Determined by Independent Central Review (ICR)
Description: PFS is defined as the time from randomization until first documentation of progression or death from any cause, whichever occurs first, as assessed by the ICR per 2008 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) guidelines with modifications for treatment-related lymphocytosis in participants with CLL and the Revised Criteria for Response for Malignant Lymphoma in participants with small lymphocytic lymphoma (SLL).
Time Frame: Up to approximately 3 years and 7 months (as of cut-off date of 07MAY2021)
Population: ITT analysis set included all enrolled participants who were assigned to a treatment group
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cohort 1: Zanubrutinib Without Del(17p): Zanubrutinib in participants with CLL without del(17p); 160 mg administered twice a day until unacceptable toxicity or disease progression
Arm/Group | Cohort 1: Bendamustine + Rituximab Without Del(17p) | Cohort 1: Zanubrutinib Without Del(17p)
Number analyzed (Participants) | 238 | 241
Months | 33.7 [28.1 to NA] — Not estimable due to low number of PFS events | NA [NA to NA] — Not estimable due to low number of PFS events
Statistical Analysis 1: Comparison: Cohort 1: Bendamustine + Rituximab Without Del(17p) vs Cohort 1: Zanubrutinib Without Del(17p); Test type: Superiority; p < 0.0001, Log Rank — One-sided; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.28 to 0.63]

2. Secondary Outcome: Cohort 1: Overall Response Rate (ORR) Between Treatment Groups as Determined by ICR
Description: ORR in Cohort 1 is defined as the percentage of participants who achieve a complete response, complete response with incomplete bone marrow recovery, partial response, or partial response with lymphocytosis, determined by the ICR.
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

3. Secondary Outcome: Pooled Cohort 1/1a: Overall Response Rate (ORR) Between Treatment Groups
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

4. Secondary Outcome: Cohort 1: Overall Survival (OS) Between Treatment Groups as Determined by the ICR
Description: OS in Cohort 1 is defined as the time from randomization to the date of death due to any reason.
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

5. Secondary Outcome: Cohort 1: Duration of Response (DOR) Between Treatment Groups as Determined by the ICR
Description: Duration of response in Cohort 1 determined using the iwCLL criteria with modification for treatment related lymphocytosis (in participants with CLL) and the Lugano Classification for non-Hodgkin lymphoma (NHL; in participants with SLL), is defined as the time from the date that criteria for response (ie, partial response with lymphocytosis [PR-L] or better) are first met to the date that disease progression is objectively documented or death, whichever occurs first.
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

6. Secondary Outcome: Pooled Cohort 1/1a: Duration of Response (DOR) Between Treatment Groups
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

7. Secondary Outcome: Cohort 1: Progression-free Survival (PFS) Between Treatment Groups Determined by Investigator Assessment (IA)
Description: PFS is defined as the time from randomization until first documentation of progression or death from any cause, whichever occurs first, as assessed by the investigator per iwCLL guidelines with modifications for treatment-related lymphocytosis in participants with CLL and the Revised Criteria for Response for Malignant Lymphoma in participants with SLL.
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

8. Secondary Outcome: Pooled Cohort 1/1a: Progression-free Survival (PFS) Between Treatment Groups Determined by Investigator Assessment (IA)
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

9. Secondary Outcome: Cohort 1: Patient-reported Outcomes as Assessed by the (European Quality Of Life 5D 5L) EQ-5D-5L Questionnaire
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

10. Secondary Outcome: Cohort 1: Patient-reported Outcomes as Assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Questionnaire.
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

11. Secondary Outcome: Cohort 2: Overall Response Rate (ORR)
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

12. Secondary Outcome: Cohort 2: Progression-free Survival (PFS)
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

13. Secondary Outcome: Cohort 2: Duration of Response (DOR)
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

14. Secondary Outcome: Cohort 3: Overall Response Rate (ORR)
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

15. Secondary Outcome: Cohort 3: Progression-free Survival (PFS)
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

16. Secondary Outcome: Cohort 3: Duration of Response (DOR)
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

17. Secondary Outcome: Cohort 3: Rate of Undetectable Minimal Residual Disease (MRD4)
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

18. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2027-09

19. Secondary Outcome: Apparent Rate of Clearance of Zanubrutinib From Plasma (CL/F)CL/F
Time Frame: Predose up to 12 hours postdose
Reporting Status: Not Posted, anticipated posting 2027-09

20. Secondary Outcome: Cohort 1 Zanubrutinib Only Arms: Area-Under-Curve From Time 0 to 12 Hours Postdose (AUC0-12)
Time Frame: Predose up to 12 hours postdose
Reporting Status: Not Posted, anticipated posting 2027-09

21. Secondary Outcome: Cohort 3: Area-Under-Curve From Time 0 to 12 Hours Postdose (AUC0-12) of Zanubrutinib
Time Frame: Predose up to 12 hours postdose
Reporting Status: Not Posted, anticipated posting 2027-09

22. Secondary Outcome: Cohort 3: Area-Under-Curve From Time 0 to 12 Hours Postdose (AUC0-12) of Zanubrutinib
Time Frame: Predose up to 12 hours postdose
Reporting Status: Not Posted, anticipated posting 2027-09

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events (AEs): Up to approximately 3 years and 7 months (as of data cut-off date of 07MAY2021)
Description: All-cause mortality is reported for all randomized participants. Serious and other AEs include participants who received at least one dose of study drug.
Arm/Group | Cohort 1: Bendamustine + Rituximab Without Del(17p) | Cohort 1: Zanubrutinib Without Del(17p) | Cohort 2: Zanubrutinib With Del(17p)
All-Cause Mortality (participants affected / at risk) | 14/238 | 16/241 | 8/111
Serious Adverse Events (participants affected / at risk) | 113/227 | 88/240 | 45/111
Other Adverse Events (participants affected / at risk) | 214/227 | 208/240 | 104/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Bendamustine + Rituximab Without Del(17p) (N=227) | Cohort 1: Zanubrutinib Without Del(17p) (N=240) | Cohort 2: Zanubrutinib With Del(17p) (N=111)
Anaemia (Blood and lymphatic system disorders) | 5 (15) | 2 (6) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 (11) | 1 (1) | 1 (1)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 4 (4) | 3 (3)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oesophageal food impaction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperpyrexia (General disorders) | 1 (2) | 0 (0) | 0 (0)
Implant site erosion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 17 (19) | 2 (2) | 2 (3)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Regenerative siderotic hepatic nodule (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abscess of salivary gland (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 8 (8) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 7 (7) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Disseminated varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
H3N2 influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis B reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Neuroborreliosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 7 (8) | 4 (5) | 6 (6)
Pneumonia chlamydial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 6 (7) | 2 (2) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tick-borne fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 1 (2) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral pericarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 (8) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
External ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Skin squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Transitional cell carcinoma urethra (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Radial nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Bladder stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteral polyp (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 2 (2)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic intramural haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Bendamustine + Rituximab Without Del(17p) (N=227) | Cohort 1: Zanubrutinib Without Del(17p) (N=240) | Cohort 2: Zanubrutinib With Del(17p) (N=111)
Anaemia (Blood and lymphatic system disorders) | 41 (65) | 11 (12) | 5 (7)
Leukopenia (Blood and lymphatic system disorders) | 7 (12) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 101 (233) | 30 (62) | 13 (28)
Thrombocytopenia (Blood and lymphatic system disorders) | 30 (62) | 8 (15) | 4 (4)
Palpitations (Cardiac disorders) | 3 (3) | 10 (10) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 2 (4) | 9 (12) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 12 (13) | 11 (16) | 9 (10)
Constipation (Gastrointestinal disorders) | 43 (49) | 24 (26) | 17 (18)
Diarrhoea (Gastrointestinal disorders) | 26 (37) | 33 (42) | 20 (24)
Dry mouth (Gastrointestinal disorders) | 9 (10) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 10 (12) | 10 (12)
Haemorrhoids (Gastrointestinal disorders) | 7 (7) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 74 (107) | 24 (30) | 18 (26)
Stomatitis (Gastrointestinal disorders) | 8 (9) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 31 (40) | 17 (23) | 8 (9)
Asthenia (General disorders) | 18 (25) | 5 (6) | 4 (6)
Chest pain (General disorders) | 2 (2) | 9 (9) | 2 (2)
Chills (General disorders) | 19 (21) | 3 (3) | 5 (6)
Fatigue (General disorders) | 36 (52) | 28 (37) | 10 (14)
Oedema peripheral (General disorders) | 16 (17) | 18 (25) | 8 (9)
Peripheral swelling (General disorders) | 6 (7) | 9 (11) | 4 (4)
Pyrexia (General disorders) | 46 (69) | 15 (15) | 6 (7)
Drug hypersensitivity (Immune system disorders) | 8 (9) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 15 (17) | 6 (6) | 3 (3)
COVID-19 (Infections and infestations) | 7 (8) | 16 (16) | 3 (5)
Cellulitis (Infections and infestations) | 2 (2) | 12 (15) | 2 (2)
Conjunctivitis (Infections and infestations) | 6 (9) | 4 (4) | 4 (7)
Herpes zoster (Infections and infestations) | 9 (9) | 5 (5) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 4 (6) | 8 (11) | 6 (6)
Nasopharyngitis (Infections and infestations) | 12 (15) | 16 (16) | 11 (13)
Oral herpes (Infections and infestations) | 7 (8) | 3 (3) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (3) | 4 (5)
Pneumonia (Infections and infestations) | 13 (14) | 8 (9) | 8 (11)
Respiratory tract infection (Infections and infestations) | 8 (9) | 7 (15) | 5 (6)
Sinusitis (Infections and infestations) | 10 (11) | 12 (12) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 27 (32) | 41 (53) | 23 (29)
Urinary tract infection (Infections and infestations) | 16 (28) | 16 (29) | 9 (11)
Contusion (Injury, poisoning and procedural complications) | 8 (8) | 46 (58) | 22 (31)
Fall (Injury, poisoning and procedural complications) | 7 (12) | 9 (11) | 9 (9)
Infusion related reaction (Injury, poisoning and procedural complications) | 39 (44) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 4 (5) | 4 (4) | 6 (7)
Alanine aminotransferase increased (Investigations) | 10 (18) | 3 (7) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 9 (12) | 3 (6) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 2 (2) | 4 (4)
Neutrophil count decreased (Investigations) | 28 (69) | 6 (14) | 7 (17)
Platelet count decreased (Investigations) | 11 (20) | 2 (2) | 4 (13)
Weight decreased (Investigations) | 7 (7) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 18 (18) | 7 (10) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 8 (13) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 4 (6) | 4 (5) | 6 (7)
Hyperuricaemia (Metabolism and nutrition disorders) | 9 (13) | 6 (7) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (26) | 4 (5) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (24) | 32 (40) | 22 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (20) | 21 (26) | 16 (19)
Bone pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 1 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 8 (10) | 7 (8)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (8) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 9 (11) | 6 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 7 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (13) | 15 (23) | 10 (11)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 9 (12) | 12 (17)
Dizziness (Nervous system disorders) | 10 (13) | 19 (21) | 8 (10)
Headache (Nervous system disorders) | 17 (19) | 26 (31) | 11 (14)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 1 (1) | 4 (4)
Sciatica (Nervous system disorders) | 4 (5) | 3 (4) | 4 (4)
Insomnia (Psychiatric disorders) | 16 (17) | 10 (11) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 8 (9) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 5 (5) | 12 (16) | 10 (12)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 3 (3) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (27) | 27 (33) | 14 (18)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 8 (8) | 11 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 12 (22) | 7 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 10 (11) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 9 (10) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (8) | 3 (3)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (8) | 6 (8)
Erythema (Skin and subcutaneous tissue disorders) | 8 (11) | 7 (8) | 3 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 18 (22) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (22) | 20 (24) | 10 (11)
Rash (Skin and subcutaneous tissue disorders) | 42 (59) | 26 (31) | 16 (19)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (12) | 8 (10) | 4 (4)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (12) | 5 (5)
Haematoma (Vascular disorders) | 1 (1) | 13 (18) | 6 (8)
Hypertension (Vascular disorders) | 19 (21) | 28 (36) | 10 (13)
Hypotension (Vascular disorders) | 21 (25) | 6 (6) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT03336333/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT03336333/SAP_001.pdf